CLINICAL TRIAL: NCT03147469
Title: The Influence of Head and Neck Position on Performance of Ambu AuraGain™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H-1704-068-844
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: General Anesthesia

STUDY DESIGN:
Intervention Model Description: AuraGain will be placed in all patients, and mechanical ventilation will be performed using a volume-controlled mode with a tidal volume of 10 ml/kg.
  The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed first for the neutral head position and then for the extended, flexed, and rotated head positions in a random order.
  Fiberoptic bronchoscopic view will be also assessed for each head and neck positions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neutral (No Intervention): After insertion of Ambu AuraGain™, the variables will be assessed at each positions including neutral, flexion, extension, right rotation under random order.
- Flexion (Experimental): After positioning the subjects' neck to flexion, the variables will be assessed.
  Interventions: Procedure: Flexion
- Extension (Experimental): After positioning the subjects' neck to extension, the variables will be assessed.
  Interventions: Procedure: Extension
- Right rotation (Experimental): After positioning the subjects' head to right rotation, the variables will be assessed.
  Interventions: Procedure: Right rotation

INTERVENTIONS:
Procedure: Flexion — After changing the position of head and neck of subjects to flexion, the variables were measured.
  Arms: Flexion
Procedure: Extension — After changing the position of head and neck of subjects to extension, the variables were measured.
  Arms: Extension
Procedure: Right rotation — After changing the position of head and neck of subjects to right flexion, the variables were measured.
  Arms: Right rotation

SUMMARY:
The influence of different head and neck positions on the effectiveness of ventilation with the Ambu AuraGain airway remains unevaluated.

This study aimed to evaluate the influence of different head and neck positions on ventilation with the AuraGain airway.

AuraGain will be placed in all patients, and mechanical ventilation will be performed using a volume-controlled mode with a tidal volume of 10 ml/kg.

The expiratory tidal volume, peak inspiratory pressure, oropharyngeal leak pressure, and ventilation score will be assessed first for the neutral head position and then for the extended, flexed, and rotated head positions in a random order.

Fiberoptic bronchoscopic view will be also assessed for each head and neck positions.

ELIGIBILITY:
Inclusion Criteria:

* Adults who were to undergo elective surgery under general anaesthesia using supraglottic airway device

Exclusion Criteria:

* Patients who had risk factor for difficult intubation
* BMI > 30kg/m2
* Emergency operation without NPO
* History of cervical spine surgery or disease
* History of esophageal operation or gastroesophageal reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 30 seconds after positioning of head and neck
  The airway pressure at which a leak sound is detected around the patient's mouth and at which the airway pressure has reached equilibrium, when the pressure-limiting valve of the anesthesia breathing system is closed and the fresh gas flow rate was fixed at 3 L/min.

SECONDARY OUTCOMES:
Peak inspiratory pressure | 30 seconds after positioning of head and neck
  Peak inspiratory pressure
Expiratory tidal volume | 30 seconds after positioning of head and neck
  Expiratory tidal volume
Ventilation score | 30 seconds after positioning of head and neck
  No leakage with an airway pressure of 15cmH2O; bilateral chest excursion with a peak inspiratory pressure of 20cmH2O; and a square-wave capnogram
Fiberoptic score | 30 seconds after positioning of head and neck
  1, vocal cords not visible; 2, vocal cords plus anterior epiglottis visible; 3, vocal cords plus posterior epiglottis visible; 4, only vocal cords visible

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided